CLINICAL TRIAL: NCT07025629
Title: Dapagliflozin for Cardio-renal Protection After ICU Discharge: A Prospective, Randomized, Double Blinded, Multicenter Study: "DAPA-ICU Trial"
Brief Title: Dapagliflozin for Cardio-renal Protection After ICU Discharge
Acronym: DAPA-ICU
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP220826
Record Dates: First submitted 2025-05-12; First posted 2025-06-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure and Chronic Kidney Disease Post-ICU
Keywords: Cardiovascular outcomes; Renal outcomes; SGLT2 inhibitors; Cardiorenal syndrome; Critical illness recovery
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: Two groups of participants will each receive different interventions.One group will receive dapagliflozin for the same amount of time that a second group will receive Placebo of dapagliflozin .
Who Masked: Participant, Investigator
Masking Description: Treatments will be conditioned and labelled by the Contract manufacturing organization AGEPS according to a list provided by an independent person and assigning a treatment arm to each treatment number.
  Randomization and treatment numbers lists are kept strictly confidential until the time of unblinding, and will not be accessible by anyone involved in the study, with the exception of the independent, unblinded statistician approving the randomization scheme; the study will be kept blinded to patients, investigators and study personnel also during the entire study period; The identification of treatment will be concealed by the use of a matching placebo to the study product that will be provided in boxes identical in packaging, labeling and appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): One tablet of dapagliflozin 10 mg will be administered once daily from randomization and for 12 months period +/- 15 days..
  Interventions: Drug: Dapagliflozin 10 MG Oral Tablet [Farxiga]
- Placebo of dapagliflozin (Placebo Comparator): One tablet of placebo of dapagliflozin 10 mg will be administered, per os, once daily from randomization and for 12 months period ± 15 days.
  Interventions: Drug: One tablet of placebo of dapagliflozin 10 mg

INTERVENTIONS:
Drug: Dapagliflozin 10 MG Oral Tablet [Farxiga] — One tablet of dapagliflozin 10 mg will be administered once daily from randomization and for 12 months period +/- 15 days..
  Arms: Dapagliflozin
Drug: One tablet of placebo of dapagliflozin 10 mg — One tablet of placebo of dapagliflozin 10 mg will be administered, per os, once daily from randomization and for 12 months period ± 15 days.
  Arms: Placebo of dapagliflozin

SUMMARY:
Several millions of patients are admitted to ICUs in Europe or USA each year. We and others, have shown that patients discharged from intensive care units (ICU) have a high incidence of cardiovascular and/or renal events and high mortality rate (22%) during the year following ICU discharge. Furthermore, a very recent meta-analysis found an excess hazard of late cardiovascular events which persists for at least 5 years following hospital discharge in sepsis survivors. Hence, many international ICU societies recommended investigating and improving post-ICU outcome with scarce guidance. We demonstrated that the proportion of ICU patients dying or presenting cardiovascular events within the year following ICU discharge is reported ~25% [2], reaching ~40% in some studies when considering patients with acute kidney injury (AKI). Plasma biomarkers at ICU discharge have good predictive value and patients with increased kidney or cardiovascular biomarkers display high risk of such events. In addition, we and others demonstrated that AKI or sub-AKI (patient not meeting the AKI definition but with an increased kidney related biomarker) could induce remote cardio-vascular injury and fibrosis, which may be involved in the poor long-term prognosis of ICU-acquired AKI. We hypothesize that strategy that prevent worsening in cardiovascular and/or renal injuries and/or in cardiovascular consequences of sub-AKI and AKI after ICU discharge improve long-term outcomes in ICU survivors. SGLT2 inhibitors are widely recognized as key drugs to protect the kidney and/or the myocardium in chronic diseases such as diabetes or heart failure. Cardio protective effect of SGLT2 inhibitors is optimal in patients with higher cardiac biomarker.

DETAILED DESCRIPTION:
Phase III study Prospective, multicenter, superiority, double-blind, randomized controlled study with two arms (1:1).

Every patient will be screened in the 48h before ICU discharge for trial inclusion and non-inclusion criteria until 72h hours after ICU discharge. After providing written informed consent, patients will be randomly assigned to receive either dapagliflozin (at a dose of 10 mg once daily) or matching placebo, in accordance with the sequestered, fixed-randomization schedule, with the use of balanced blocks to ensure an approximate 1:1 ratio of the two regimens for one year.

Four visits are planned, one at inclusion (V0), one at 6 months (V1), one at the end of the treatment (V2 at one year), one 6 weeks after the end of the treatment (V3, end of the study) and two phone calls at 3 (Phone call 1) and 9 months (phone call 2).

At 6 months (V1) and at 12 months (V2) visits, a clinical exam and biological analysis will be performed at hospital (i.e., HbA1c, glucose level, ionogram, NT-proBNP or BNP, serum creatinine, hematocrit and pregnancy urinary test) by anesthesiologists, cardiologists or nephrologists, to assess primary and secondary endpoints, including eGFR.

At 12 months + 6 weeks (V3) visit, a clinical exam and biological analysis will be performed at hospital (i.e., glucose level, NT-proBNP or BNP, serum creatinine) by anesthesiologists, cardiologists or nephrologists, to assess primary and secondary endpoints, including eGFR.

The phone calls, at 3 and 9 months, will be made by the designated persons and respecting the confidentiality and security of the data collected.

At inclusion (V0) and at 6 months (V1) the treatment will be deliver for the next 6 months. At 6 months (V1), the patient will pick up his treatment at the hospital.

Primary endpoints will be assessed at 6 and 12 months visit and phone calls (3 and 9 months).

Secondary endpoints will be assessed at each visit and phone calls (3, 6, 9, 12 and 12 + 6 weeks).

eGFR (glomerular filtration rate) will be assessed only at 6, 12 months and 12 + 6 weeks. The eGFR (glomerular filtration rate) will not be assessed at phone calls.

At each visit and phone calls, adverse events and severe adverse events will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age >or= 18 years
* Mechanical ventilation and/or vasopressors/inotropes for more than 24h during ICU stay
* Patients ready to be discharged from ICU according to physician in charge
* Inform consent form signed by the patient
* NT-proBNP greater than 800 ng/L or BNP > 90 ng/L and/or Estimated glomerular filtration rate (eGFR) between 25ml/min/1.73m² and 90ml/min/1.73m² of body-surface area (CKD-EPI formula) at inclusion.

Exclusion Criteria:

* Pregnancy
* Ability to become pregnant and refusal to use effective contraception during all study treatment Women of childbearing potential (WOCBP)** must agree to use adequate contraception according to Recommendations related to contraception and pregnancy testing in clinical trials, by Clinical Trial Facilitation Group (CTFG).

The inclusion of WOCBP requires use of a highly effective contraceptive measure :

* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

  * oral
  * intravaginal
  * transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation

  * oral
  * injectable
  * implantable
* intrauterine device (IUD)
* intrauterine hormone-releasing system ( IUS)
* bilateral tubal occlusion
* vasectomised partner
* sexual abstinence

The above mentioned risk mitigation measures (contraception) should be maintained during treatment and until the end of relevant systemic exposure.

** a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

* Breast feeding
* Known hypersensitivity to dapagliflozin or any of the excipients
* Patients treated with dapagliflozin before ICU admission
* Patients with severe cirrhosis (Child-Pugh C)
* Patients who admitted or who developed during their ICU stay a urinary tract infection or a perineal infection and patients at risk of skin infection near the perineum (e.g., a sacral pressure ulcer)
* Estimated glomerular filtration rate (eGFR) below 25 ml per minute per 1.73 m2 of body-surface area (CKD -EPI formula).
* Patient for whom treatment with Dapagliflozine is strongly recommended according to recent international guidelines:

  * patients with type 2 diabetes mellitus adults for whom the treatment is inadequately controlled as an adjunct to diet and exercise: either as monotherapy when metformin is considered inappropriate due to inadequate tolerance, or in addition to other medications for the treatment of type 2 diabetes,
  * symptomatic chronic heart failure with reduced or preserved left ventricular ejection fraction,
  * chronic kidney disease, in addition to standard therapy with a glomerular filtration rate (GFR) between 25 and 75 mL/min/1.73m² and a urinary albumin-to-creatinine ratio (ACR) between 200 and 5000 mg/g and treated for at least 4 weeks with an ACE inhibitor or angiotensin 2 receptor blocker (ARB II or sartan).
* Patient without national health insurance, and patient on AME (state medical aid)
* Persons deprived of liberty by a judicial or administrative decision
* Participation in other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Within the year after randomization
Unscheduled hospital hospitalization for heart failure | Within the year after randomization
  All potential hospitalizations for heart failure should be recorded in the eCRF and submitted to adjudication. The Clinical Event Adjudication (CEA) committee members will adjudicate the events as specified in the (CEA) Charter.
Decrease of eGFR by more than 50% from ICU discharge and/or end stage kidney disease defined as an eGFR<15ml/min/1.73m² and/or initiation of renal replacement therapy and/or kidney transplantation | Within the year after randomization
  Dialysis, eGFR events (<15 mL/min/1.73m²; ≥50% decline in eGFR) will be recorded in the eCRF and submitted for adjudication.
  eGFR baseline is defined as the local laboratory value at inclusion visit. The eGFR will be calculated using CKD-EPI equation without race coefficient [87, 88].

SECONDARY OUTCOMES:
Unscheduled hospital hospitalization for acute heart failure | Within the year after randomization
Unscheduled hospital hospitalization for stroke | Within the year after randomization
Unscheduled hospital hospitalization for acute coronary syndrome | Within the year after randomization
Occurrence of severe chronic kidney disease | Within the year after randomization
  Defined as eGFR <30 ml/min/1.73m2
• Decrease of estimated glomerular filtration rate of more than 50% from baseline | Within the year after randomization
New episode of acute kidney injury (according to the KDIGO criteria) requiring hospitalization | Within the year after randomization
Occurrence of end stage kidney disease defined (eGFR<15ml/min/1.73m2) and/or initiation of renal replacement therapy and/or kidney transplantation | Within the year after randomization
Change in NT-proBNP (pg/mL) from baseline to end of study | Between 12 months (end of treatment) and 12 months + 6 weeks (end of study)
Occurrence of cardiovascular events | Within the year after randomization
  The participants sites should record potential strokes and transit ischemic attacks (TIAs) in the eCRF and submit for adjudication. The CEA committee members will adjudicate all potential cerebrovascular events to decide if they qualify as stroke according to the criteria defined in the CEA charter
Occurrence of renal events | Within the year of treatment
Urinary tract infection | Within the year after randomization
  All potential events of urinary tract infection will be recorded in the eCRF and submitted to the CEA.
Necrotizing fasciitis | Within the year after randomization
  All potential events of necrotizing fasciitis will be recorded in the eCRF and submitted to the CEA.
Symptomatic ketoacidosis | Within the year after randomization
  This outcome is defined as Arterial pH <7.3 and Ketone-positive urine and Anion gap >10 mEq/L and Drowsy, stupor or coma All potential events of ketoacidosis will be recorded in the eCRF and submitted to the CEA.
Major hypoglycaemia | Within the year after randomization
  This outcome is defined as gycemia<3 mmol/l) and any episode of hypoglycemia for which assistance was needed, all potential major hypoglycaemia will be recorded in the eCRF and submitted to the CEA.
Death of any cause | Within the year after randomization
Change in BNP (pg/mL) from baseline to end of study | Between 12 months (end of treatment) and 12 months + 6 weeks (end of study)
Change in estimated glomerular filtration rate (eGFR, mL/min/1.73 m²) from baseline to end of study" | Between 12 months (end of treatment) and 12 months + 6 weeks (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, MD-PHD, Principal Investigator — APHP; François DEPRET, MD-PHD, Study Chair — APHP
Locations (2):
- France (2):
  - Hospital Saint Louis, Paris
  - Saint Louis Hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared. The data will be anonymized to protect participants' privacy. Researchers may request access to the data by contacting the Steering Committee, which will review the request within two months. The data will be available one year after publication.
Time Frame: The data will be available one year after publication, for 5 years

REFERENCES:
- [Background] Sano M, Goto S. Possible Mechanism of Hematocrit Elevation by Sodium Glucose Cotransporter 2 Inhibitors and Associated Beneficial Renal and Cardiovascular Effects. Circulation. 2019 Apr 23;139(17):1985-1987. doi: 10.1161/CIRCULATIONAHA.118.038881. No abstract available. PMID 31009585
- [Background] Chang YK, Choi H, Jeong JY, Na KR, Lee KW, Lim BJ, Choi DE. Dapagliflozin, SGLT2 Inhibitor, Attenuates Renal Ischemia-Reperfusion Injury. PLoS One. 2016 Jul 8;11(7):e0158810. doi: 10.1371/journal.pone.0158810. eCollection 2016. PMID 27391020
- [Background] Zelniker TA, Wiviott SD, Raz I, Im K, Goodrich EL, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Furtado RHM, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Sabatine MS. SGLT2 inhibitors for primary and secondary prevention of cardiovascular and renal outcomes in type 2 diabetes: a systematic review and meta-analysis of cardiovascular outcome trials. Lancet. 2019 Jan 5;393(10166):31-39. doi: 10.1016/S0140-6736(18)32590-X. Epub 2018 Nov 10. PMID 30424892
- [Background] Zannad F, Ferreira JP, Pocock SJ, Anker SD, Butler J, Filippatos G, Brueckmann M, Ofstad AP, Pfarr E, Jamal W, Packer M. SGLT2 inhibitors in patients with heart failure with reduced ejection fraction: a meta-analysis of the EMPEROR-Reduced and DAPA-HF trials. Lancet. 2020 Sep 19;396(10254):819-829. doi: 10.1016/S0140-6736(20)31824-9. Epub 2020 Aug 30. PMID 32877652
- [Background] Depret F, Hollinger A, Cariou A, Deye N, Vieillard-Baron A, Fournier MC, Jaber S, Damoisel C, Lu Q, Monnet X, Rennuit I, Darmon M, Leone M, Guidet B, Sonneville R, Montravers P, Pili-Floury S, Lefrant JY, Duranteau J, Laterre PF, Brechot N, Oueslati H, Cholley B, Struck J, Hartmann O, Mebazaa A, Gayat E, Legrand M. Incidence and Outcome of Subclinical Acute Kidney Injury Using penKid in Critically Ill Patients. Am J Respir Crit Care Med. 2020 Sep 15;202(6):822-829. doi: 10.1164/rccm.201910-1950OC. PMID 32516543
- [Background] Legrand M, Rossignol P. Cardiovascular Consequences of Acute Kidney Injury. N Engl J Med. 2020 Jun 4;382(23):2238-2247. doi: 10.1056/NEJMra1916393. No abstract available. PMID 32492305
- [Background] Gayat E, Cariou A, Deye N, Vieillard-Baron A, Jaber S, Damoisel C, Lu Q, Monnet X, Rennuit I, Azoulay E, Leone M, Oueslati H, Guidet B, Friedman D, Tesniere A, Sonneville R, Montravers P, Pili-Floury S, Lefrant JY, Duranteau J, Laterre PF, Brechot N, Chevreul K, Michel M, Cholley B, Legrand M, Launay JM, Vicaut E, Singer M, Resche-Rigon M, Mebazaa A. Determinants of long-term outcome in ICU survivors: results from the FROG-ICU study. Crit Care. 2018 Jan 18;22(1):8. doi: 10.1186/s13054-017-1922-8. PMID 29347987
- [Background] Arrigo M, Feliot E, Gayat E, Mebazaa A. Cardiovascular events after ICU discharge in patients with new-onset atrial fibrillation: A report from the FROG-ICU study. Int J Cardiol. 2018 Nov 1;270:203. doi: 10.1016/j.ijcard.2018.07.080. Epub 2018 Jul 20. No abstract available. PMID 30045823